CLINICAL TRIAL: NCT01851031
Title: A New Surgical Approach to Treat Medial or Low Condylar Fractures:The Minor Parotid Anterior Approach
Brief Title: A New Surgical Approach to Treat Medial or Low Condylar Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China College of Stomatology (Other)
Responsible Party: Principal Investigator, Hou Jia, Principal Investigator, West China College of Stomatology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: houjia
Record Dates: First submitted 2013-04-27; First posted 2013-05-10 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Fracture of Condylar Process
Keywords: medial or low condylar fractures; the minor parotid anterior approach; the retromandibular approach

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the minor approach group (Experimental): Thirty-six patients (the minor parotid anterior approach group) were treated with minor parotid anterior approach
  Interventions: Procedure: the minor approach
- control group (Other): 24 patients (control group) were treated with the retromandibular approach
  Interventions: Procedure: the minor approach

INTERVENTIONS:
Procedure: the minor approach — Thirty-six patients (the minor approach group) were treated with minor parotid anterior approach
  Other Names: the minor parotid anterior approach

SUMMARY:
The aim of the study was to compare the new approach and the retromandibular approach, so that the therapeutic effect and the advantages of the new approach would be clear.

DETAILED DESCRIPTION:
Sixty patients (72 sides) with medial or low condylar fractures were treated with surgical intervention. Thirty-six patients (42 sides) were treated with minor parotid anterior approach, and the other 24 patients (30 sides) were treated with retromandibular approach. The data about the operations and complications were recorded. The follow-up periods were 3-12 months.

ELIGIBILITY:
Inclusion Criteria:

* (1)clinical and imaging diagnosis of medial or low condylar fractures
* (2)bone fragments that were obviously dislocated, that affected patients appearance and function, requiring surgical intervention
* (3)no previous surgical treatment

Exclusion Criteria:

* (1)medial or low condylar fractures without obvious displacement
* (2)patients who had previously undergone unsuccessful surgery
* (3)the surgical site had traumatic scar, so the approach could be carried out on the original incision

Ages: 5 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2009-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
the number of participants with facial nerve injury | from 3 months to 1 year after surgery
  to explore whether the minor parotid anterior approach could prevent facial nerve injury.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Hou, DMD, Study Chair — West China College of Stomatology
Locations (1):
- West China College of Stomatology, Chengdu, Sichuan, China

REFERENCES:
- [Result] Tang W, Gao C, Long J, Lin Y, Wang H, Liu L, Tian W. Application of modified retromandibular approach indirectly from the anterior edge of the parotid gland in the surgical treatment of condylar fracture. J Oral Maxillofac Surg. 2009 Mar;67(3):552-8. doi: 10.1016/j.joms.2008.06.066. PMID 19231779
- [Derived] Hou J, Chen L, Wang T, Jing W, Tang W, Long J, Tian W, Liu L. A new surgical approach to treat medial or low condylar fractures: the minor parotid anterior approach. Oral Surg Oral Med Oral Pathol Oral Radiol. 2014 Mar;117(3):283-8. doi: 10.1016/j.oooo.2013.11.491. Epub 2013 Nov 18. PMID 24405647